CLINICAL TRIAL: NCT05803161
Title: A Randomized, Double-blind, Dose-exploration, Parallel-controlled, Multicenter Phase II Clinical Study of Congrong Runtong Oral Liquid in the Treatment of Functional Constipation (Yang-deficiency Type)
Brief Title: Congrong Runtong Oral Liquid in the Treatment of Functional Constipation (Yang-deficiency Type)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, zhangshengsheng, Principal Investigator, Beijing Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KANION-CRRT-2022
Record Dates: First submitted 2023-03-26; First posted 2023-04-07 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Functional Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Congrong Runtong oral liquid high-dose group (Experimental): Congrong Runtong oral liquid, 2 bottles (1g herb content per bottle) per dose, three times a day
  Interventions: Drug: Congrong Runtong oral liquid
- Congrong Runtong oral liquid low-dose group (Experimental): Congrong Runtong oral liquid, 2 bottles (0.5g herb content per bottle) per dose, three times a day
  Interventions: Drug: Congrong Runtong oral liquid
- Placebo group (Placebo Comparator): Congrong Runtong oral liquid, 2 bottles (0g herb content per bottle) per dose, three times a day
  Interventions: Drug: Placental Congrong Runtong oral liquid

INTERVENTIONS:
Drug: Congrong Runtong oral liquid — Congrong Runtong oral liquid：component "total glycosides of Cistanche" extracted and refined from the traditional Chinese medicine Cistanche deserticola
  Arms: Congrong Runtong oral liquid high-dose group; Congrong Runtong oral liquid low-dose group
Drug: Placental Congrong Runtong oral liquid — Placental Congrong Runtong oral liquid
  Arms: Placebo group

SUMMARY:
Using a placebo as a control, this study aims to preliminarily evaluate the clinical efficacy of Congrong Runtong oral liquid for the treatment of functional constipation (Yang-deficiency type), explore the optimal dosage of Congrong Runtong oral liquid for functional constipation (Yang-deficiency type) to provide a basis for dosage selection in Phase III clinical trials, and observe the safety of clinical use of Congrong Runtong oral liquid.

ELIGIBILITY:
Inclusion Criteria:

1. Meets the Rome IV diagnostic criteria for functional constipation;
2. Meets the TCM diagnostic criteria for Yang-deficiency type constipation;
3. Aged between 18 and 70 years (inclusive);
4. Has undergone colonoscopy and has been diagnosed with either no abnormalities or non-adenomatous polyps (size not exceeding 0.5 cm, no more than 3) or has undergone polypectomy for more than 1 month and the pathological examination confirms no high-grade intraepithelial neoplasia within 12 months of colonoscopy examination in a tertiary grade A hospital
5. Less than 3 complete spontaneous bowel movements per week during the 2-week run-in period;
6. Voluntarily participates in the trial and signs an informed consent form.

Exclusion Criteria:

1. Patients with constipation caused by organic lesions of the rectum or colon (such as tumors, inflammatory bowel disease, anal fissure, intestinal adhesions, intestinal tuberculosis) leading to intestinal stenosis;
2. Patients with constipation caused by other systemic organic diseases, such as congenital megacolon, neurological disorders (such as autonomic neuropathy, cerebrovascular disease, etc.), mental disorders, metabolic endocrine disorders (such as hypothyroidism, diabetes mellitus with fasting blood glucose > 8.6mmol/L or with complications), muscular diseases (such as amyloidosis, dermatomyositis), etc.;
3. Patients whose drug-induced constipation cannot be ruled out by the investigators；
4. Patients with alarm signs judged by the investigator and unable to exclude malignant lesions by colonoscopy in the past three months;
5. ALT or AST ≥ 1.5 times the upper limit of the normal value, or Scr > upper limit of the normal value;
6. Patients allergic to the composition of the ingredients of the Cenruong Runtong oral solution or bisacodyl;
7. Pregnant or breastfeeding women, or women planning to become pregnant;
8. Patients who have participated in other clinical trials in the past 3 months;
9. Other situations judged by the investigator as inappropriate for participation in this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Complete Spontaneous Bowel Movement (CSBM) response rate within 8 weeks of treatment | Examination will be performed after 8 weeks of treatment.
  CSBM response: the patient meets the CSBM weekly response at least 50% of the time during the weeks of drug treatment (e.g., 4/8 weeks).
  Weekly response: The patient has at least 3 CSBMs per week and has an increase of at least one CSBM compared to baseline, which is considered a weekly response.
  Overall CSBM response rate = CSBM response number / total observed number of people × 100%"

SECONDARY OUTCOMES:
The occurrence of CSBM within the first 24 hours of starting treatment | Evaluation will be performed after 24 hours of treatment.
  Calculate the number of CSBM during the first 24 hours of treatment
Changes in the number of bowel movements (BM)compared to baseline at 2, 4, 6, and 8 weeks | Evaluation will be performed at baseline and after2，4，6，8 weeks of treatment.
  The patient recorded the number of BMs every day using a diary card, and the weekly number of BMs was the total of the seven days
Changes in the number of spontaneous bowel movements (SBM)compared to baseline at 2, 4, 6, and 8 weeks | Evaluation will be performed at baseline and after2，4，6，8 weeks of treatment.
  The patient recorded the number of SBMs every day using a diary card, and the weekly number of SBMs was the total of the seven days
Changes in the fecal characteristics score (using the Bristol Stool Form Scale) compared to baseline at 2, 4, 6, and 8 weeks | Evaluation will be performed at baseline and after2，4，6，8 weeks of treatment.
  Bristol Stool Form Scale： Type 1 Separate hard lumps, like nuts. Type 2 Sausage-shaped but lumpy. Type 3 Like a sausage or snake but with cracks on its surface. Type 4 Like a sausage or snake, smooth and soft. Type 5 Soft blobs with clear-cut edges. Type 6 Fluffy pieces with ragged edges, a mushy stool.
  Type 7 Watery, no solid pieces. The 1-7 types correspond to scores of 1-7 respectively.
Changes in the degree of difficulty in passing stools score (using the Likert scale) compared to baseline at 2, 4, 6, and 8 weeks | Evaluation will be performed at baseline and after2，4，6，8 weeks of treatment.
  The Patient Assessment of Constipation Symptoms (PAC-SYM) questionnaire uses a Likert scale grading system for rating the severity of constipation symptoms, which is divided into five levels of severity: 0, 1, 2, 3, and 4.
The average number of CSBMs per week | Examination will be performed after 8 weeks of treatment.
  The average number of CSBMs per week is calculated by dividing the total number of CSBMs during the observation period by the number of observation weeks (8 weeks)
The average number of SBMs per week | Examination will be performed after 8 weeks of treatment.
  The average number of SBMs per week is calculated by dividing the total number of SBMs during the observation period by the number of observation weeks (8 weeks)
The average fecal characteristic score per week (using the Bristol Stool Chart) | Examination will be performed after 8 weeks of treatment.
  The stool consistency score for each week is calculated by dividing the sum of all stool consistency scores for that week by the total number of bowel movements during that week.The average stool consistency score per week is calculated by dividing the sum of all weekly stool consistency scores by the number of observation weeks (8 weeks).
The use of rescue medication | Examination will be performed after 8 weeks of treatment.
  Calculate the total number of rescue medication doses taken during the treatment period
The changes in TCM syndrome scores compared to baseline at 4 and 8 weeks of treatment | Examination will be performed at baseline and after 4,8 weeks of treatment.
  The TCM syndrome score of functional constipation consists of 5 questions, and the total scores are ranging from 0 to 24 with higher scores indicating more severe disease.
Changes in the Patient Assessment of Constipation Quality of Life (PAC-QOL) score compared to baseline at 4 and 8 weeks of treatment | Examination will be performed at baseline and after4，8 weeks of treatment.
  Calculate the total PAC-QOL score and the change in scores for the physiological, psychosocial, worries, and satisfaction domains compared to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Hospital of Traditional Chinese Medicine, Capital Medical University, Beijing, Dongcheng, China

IPD SHARING:
Plan to Share IPD: No